CLINICAL TRIAL: NCT05163951
Title: Effectiveness and Safety of Trabeculectomy and Peripheral Iridectomy Plus Goniotomy in Advanced Primary Angle-closure Glaucoma: a Multicenter Non-inferiority Randomized Controlled Trial
Brief Title: Trabeculectomy Versus Peripheral Iridectomy Plus Goniotomy in Advanced PACG
Acronym: TVG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other); First Hospital of Shijiazhuang City (Other); West China Hospital (Other); Chongqing Medical University (Other); Handan City Eye Hospital (Unknown); People's Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Director of Clinical Research Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021KYPJ191
Record Dates: First submitted 2021-11-25; First posted 2021-12-20 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Primary Angle Closure Glaucoma
Keywords: angle closure; glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure; Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Intervention Model Description: multicenter, parallel, open, non-inferior randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trabeculectomy (Active Comparator): Forty-four patients with advanced primary angle closure glaucoma will receive trabeculectomy.
  Interventions: Procedure: Trabeculectomy
- SPI+GSL+GT (Experimental): Forty-four patients with advanced primary angle closure glaucoma will receive surgical peripheral iridectomy (SPI) combined with goniosynechialysis (GSL) and goniotomy (GT).
  Interventions: Procedure: SPI+GSL+GT

INTERVENTIONS:
Procedure: Trabeculectomy — trabeculectomy
  Arms: Trabeculectomy
Procedure: SPI+GSL+GT — Peripheral iridectomy (SPI) combined with goniosynechialysis (GSL) and goniotomy (GT)
  Arms: SPI+GSL+GT

SUMMARY:
A multicenter, parallel, open, non-inferior randomized controlled trial is conducted to compare the effectiveness and safety of trabeculectomy and peripheral iridectomy plus goniotomy (TVG) in the treatment of advanced primary angle closure glaucoma with no or mild cataracts.

DETAILED DESCRIPTION:
Primary angle-closure glaucoma (PACG) has a high prevalence and blinding rate in China. The routine first-line treatment of advanced PACG is trabeculectomy, especially in those without cataract. However, due to surgery complications and exhausting post-surgery caring, traditional trabeculectomy is not an ideal choice in clinical practice, particularly in patients with high risk of complications such as younger age and shorter axial length. Peripheral iridectomy (SPI) plus intraocular pressure (IOP)-lowering medications is an alternative.

Minimally invasive glaucoma surgery (MIGS) has recently showed its safety and effectiveness in the treatment of PACG, usually combined with cataract surgery, goniosynechialysis (GSL) and goniotomy(GT). The safety and effectiveness of phacoemulsification and intraocular lens implantation (PEI)+GSL+GT in advanced PACG with cataract has been conducted (clinical trials.gov, NCT04878458). It is valuable to explore the safety and efficacy of SPI+GSL+GT in these PACG patients with no or mild cataracts.

Therefore, this study intends to conduct a multicenter, non-inferior randomized controlled clinical trial to compare the effectiveness and safety of trabeculectomy versus SPI+GSL+GT in advanced PACG with no or mild cataracts.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-80 years.
2. Eyes diagnosed with advanced PACG who meet following criteria a, b, and c; or a, b, and d:

   1. PAS: ≥180° range, including nasal and inferior quadrants;
   2. IOP >21 mmHg with or without anti-glaucoma medications (the medications include the maximally tolerated medications), taken with the Goldmann applanation tonometer;
   3. Glaucomatous optic neuropathy (cup-to-disc [C/D] ratio ≥0.7, C/D asymmetry >0.2, or rim width at the superior and inferior temporal areas <0.1 of the vertical diameters of the optic disc);
   4. Glaucomatous visual field defects (nasal step, arcuate scotoma, and paracentral scotoma on a reliable Humphrey analyzer and a mean deviation of ≤-12 dB).
3. No or mild cataracts and uncorrected visual acuity of ≥0.63 (Early Treatment Diabetic Retinopathy Study chart);
4. Axial length of ≥20 mm.

Exclusion Criteria:

1. History of ocular surgery or trauma.
2. Retinal disease that influences the collection of ocular parameters or other types of glaucoma, including open-angle glaucoma, secondary angle-closure glaucoma, steroidal glaucoma, angle recession glaucoma, neovascular glaucoma, nanophthalmos, and pseudoexfoliation syndrome.
3. Monophthalmia (best-corrected visual acuity of <0.01 in the non-study eye).
4. An International Standardized Ratio of >3.0, for patients receiving warfarin or anticoagulant therapy before surgery.
5. Patients with serious systemic diseases.
6. Pregnant or lactating women.

If both eyes are eligible for the study, the eye with the worse visual field or optic nerve will be included.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure at postoperative 12 months | Postoperative 12 month
  Intraocular pressure after surgery using Goldmann or non-contact tonometer.

SECONDARY OUTCOMES:
Cumulative success rate of surgery | Postoperative 12, 24, 36 months
  Cumulative success rate of surgery is defined as :
  (i) Complete success is defined as the postoperative intraocular pressure between 5 and 18 mmHg, and 20% reduction from baseline without anti-glaucoma medications.
  (ii) Qualified success is defined as the postoperative intraocular pressure between 5 and 18 mmHg, and 20% reduction from baseline with anti-glaucoma medications.
Intraoperative and postoperative complications | Postoperative 0, 1, 7 days, and 1, 3, 6, 12, 18, 24, 30, 36 months
  Intraoperative and postoperative complications, such as shallow anterior chamber, malignant glaucoma, hyphema, persistent hypotony, corneal endothelium decompensation, endophthalmitis, and bleb-related complications.
The numbers of anti-glaucoma medications | Postoperative 0, 1, 7 days, and 1, 3, 6, 12, 18, 24, 30, 36 months
  Numbers of anti-glaucoma medications.

OTHER OUTCOMES:
Visual acuity | Postoperative 0, 1, 7 days, and 1, 3, 6, 12, 18, 24, 30, 36 months
  Uncorrected and best corrected visual acuity will be documented using ETDRS chart.
The degree of peripheral anterior synechia | Postoperative 0, 3, 12, 24, 36 months
  The peripheral anterior synechia is checked using gonioscopy. Range from 0-360° will be documented.
Corneal endothelial cell counting | Postoperative 0,12, 24, 36 months
  Corneal endothelial cell counting will be documented using specular microscope.
Visual field | Postoperative 0,6,12, 24, 36 months
  Visual field will be performed using Humphrey analyzer, in which parameters of mean deviation (MD), pattern standard deviation (PSD) will be documented.
Optic nerve head morphology | Postoperative 0,12, 24, 36 months
  Optic nerve head morphology will be derived from optical coherence tomography (Cirrus 5000, Carl Zeiss Meditec, USA or Heidelberg OCT, SPECTRALIS OCT, Heidelberg, Germany).
Retinal thickness | Postoperative 0,12, 24, 36 months
  Retinal thickness will be derived from optical coherence tomography (Cirrus 5000, Carl Zeiss Meditec, USA or Heidelberg OCT, SPECTRALIS OCT, Heidelberg, Germany).
The quality of life | Postoperative 0,12, 24, 36 months
  Quality of life will be measured with EQ-5D-5L questionnaire.
Filtering bleb classification | Postoperative 3, 12, 24, 36 months
  Filtering bleb classification using the Indiana Bleb Appearance Grading Scale, including height, width, extent, vascularity, and Seidel test.
Surgical time | Postoperative 1 day
  Surgical time will be documented.
Surgical cost | Postoperative 1 day
  Surgical cost will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Xiulan Zhang, MD. PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Husain R, Do T, Lai J, Kitnarong N, Nongpiur ME, Perera SA, Ho CL, Lim SK, Aung T. Efficacy of Phacoemulsification Alone vs Phacoemulsification With Goniosynechialysis in Patients With Primary Angle-Closure Disease: A Randomized Clinical Trial. JAMA Ophthalmol. 2019 Oct 1;137(10):1107-1113. doi: 10.1001/jamaophthalmol.2019.2493. PMID 31294768
- [Result] Barry M, Alahmadi MW, Alahmadi M, AlMuzaini A, AlMohammadi M. The Safety of the Kahook Dual Blade in the Surgical Treatment of Glaucoma. Cureus. 2020 Jan 16;12(1):e6682. doi: 10.7759/cureus.6682. PMID 31976190
- [Result] Tanito M, Sugihara K, Tsutsui A, Hara K, Manabe K, Matsuoka Y. Midterm Results of Microhook ab Interno Trabeculotomy in Initial 560 Eyes with Glaucoma. J Clin Med. 2021 Feb 17;10(4):814. doi: 10.3390/jcm10040814. PMID 33671386
- [Result] Grover DS, Smith O, Fellman RL, Godfrey DG, Gupta A, Montes de Oca I, Feuer WJ. Gonioscopy-assisted Transluminal Trabeculotomy: An Ab Interno Circumferential Trabeculotomy: 24 Months Follow-up. J Glaucoma. 2018 May;27(5):393-401. doi: 10.1097/IJG.0000000000000956. PMID 29613978
- [Result] Dorairaj S, Tam MD, Balasubramani GK. Two-Year Clinical Outcomes of Combined Phacoemulsification, Goniosynechialysis, and Excisional Goniotomy For Angle-Closure Glaucoma. Asia Pac J Ophthalmol (Phila). 2020 Oct 6;10(2):183-187. doi: 10.1097/APO.0000000000000321. PMID 33031110
- [Result] Tham CC, Kwong YY, Baig N, Leung DY, Li FC, Lam DS. Phacoemulsification versus trabeculectomy in medically uncontrolled chronic angle-closure glaucoma without cataract. Ophthalmology. 2013 Jan;120(1):62-7. doi: 10.1016/j.ophtha.2012.07.021. Epub 2012 Sep 15. PMID 22986111
- [Result] Gedde SJ, Feuer WJ, Lim KS, Barton K, Goyal S, Ahmed IIK, Brandt JD; Primary Tube Versus Trabeculectomy Study Group. Treatment Outcomes in the Primary Tube Versus Trabeculectomy Study after 3 Years of Follow-up. Ophthalmology. 2020 Mar;127(3):333-345. doi: 10.1016/j.ophtha.2019.10.002. Epub 2019 Oct 9. PMID 31727428
- [Derived] Lin F, Lv A, Li F, Song Y, Xie L, Zhu X, Tang L, Zhang Y, Huang J, Tang G, Zhang H, Lu L, Xiao M, Xu J, Nie X, Liao M, Yang Y, Gao K, Yuan H, Song W, Zuo C, Lu P, Yan X, Zhou F, Wang Z, Jin L, Peng Y, Chen W, Barton K, Park KH, Aung T, Lam DSC, Weinreb RN, Wang N, Tham CC, Fan S, Zhang X; TVG study group. Peripheral Iridectomy With Goniosynechialysis and Goniotomy vs Trabeculectomy for Advanced PACG: A Randomized Clinical Trial. JAMA Ophthalmol. 2025 Jun 1;143(6):472-479. doi: 10.1001/jamaophthalmol.2025.0757. PMID 40244579
- [Derived] Gao X, Lv A, Lin F, Lu P, Zhang Y, Song W, Zhu X, Zhang H, Liao M, Song Y, Hu K, Zhang Y, Peng Y, Tang L, Yuan H, Xie L, Tang G, Nie X, Jin L, Fan S, Zhang X; TVG study group. Efficacy and safety of trabeculectomy versus peripheral iridectomy plus goniotomy in advanced primary angle-closure glaucoma: study protocol for a multicentre, non-inferiority, randomised controlled trial (the TVG study). BMJ Open. 2022 Jul 4;12(7):e062441. doi: 10.1136/bmjopen-2022-062441. PMID 35788072